CLINICAL TRIAL: NCT01847859
Title: Feasibility and Reliability of Routine Ultrasound Examination Performed by Nurses in Cardiothoracic Post-operative Patients
Brief Title: Pocket-size Ultrasound by Nurses in Cardiothoracic Post-operative Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LH-2013-2; Spl postop hjerte (Other: Levanger Hospital)
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Cardiothoracic Surgery
Keywords: Cardiothoracic surgery; Post-operative; Nurses; Cardiac; Echocardiography; Pocket-size; Hand-held
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound performed by nurses (Experimental): Focused examination of the pleural and pericardial cavity. Cardiologists perform reference ultrasound examinations.
  Interventions: Procedure: Ultrasound examination by nurses

INTERVENTIONS:
Procedure: Ultrasound examination by nurses — Focused examination of the pleural space and inferior vena cava.Reference method: Cardiologists performed ultrasound examinations.
  Other Names: Ultrasound

SUMMARY:
The investigators aim to study the feasibility and reliability of pocket-size diagnostic ultrasound examinations performed by nurses of postoperative patients who have underwent cardiothoracic surgery in a cardiac unit.

DETAILED DESCRIPTION:
Patient inclusion: Post-operative cardiothoracic surgery patients transferred to a cardiac unit. All such patients are eligible for inclusion if they consent to participate in the study. No other exclusion criteria other than not willing/able to give their consent. Only postoperative patients will be included.

Study population: Approximately 50 patients

Intervention: All participants will undergo careful medical history, physical examination and blood tests led by residents. All patients will routinely be examined with ultrasound by nurses trained in ultrasound examinations of the pleural space and the pericardium and a complete high-end echocardiography including assessment of both pleural cavities and the pericardial space will be performed in all by cardiologists.

Statistics and results: Feasibility and reliability will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative cardiothoracic patients admitted to the cardiac unit at the local hospital

Exclusion Criteria:

* Not able or not willing to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Feasibility and reliability | 0 days
  Feasibility: Proportion of patients where the pleural and pericardial cavitis can be assessed and interpreted by ultrasound performed by nurses compared with cardiologists.
Reliability | 0 days
  Validation of ultrasound examinations and interpretation of the pleural and pericardial cavities by nurses compared with cardiologists as reference.

SECONDARY OUTCOMES:
Time use | 0 days
  Comparison of the time use of ultrasound examinations of the pleural and pericardial cavities when examinations are performed by nurses and cardiologists, respectively.

OTHER OUTCOMES:
Clinical impact | 0 days and 30 days
  Clinical influence of detection/assessment of pleural and pericardial effusion by ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of medicine, Levanger Hospital, Nord-Trøndelag Health Trust, Levanger, Norway

REFERENCES:
- [Derived] Graven T, Wahba A, Hammer AM, Sagen O, Olsen O, Skjetne K, Kleinau JO, Dalen H. Focused ultrasound of the pleural cavities and the pericardium by nurses after cardiac surgery. Scand Cardiovasc J. 2015 Feb;49(1):56-63. doi: 10.3109/14017431.2015.1009383. Epub 2015 Feb 6. PMID 25611808